CLINICAL TRIAL: NCT03351842
Title: A PHASE II STUDY Of ADJUVANT CHEMOTHERAPY After SURGERY For STAGE I Lung ADENOCARCINOMA PATIENTS With MICROPAPILLARY COMPONENT More Than Or EQUAL To 20%
Brief Title: Surgery With or Without Chemotherapy for Stage I NSCLC With Micropapillary Component ≥ 20%
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Gening Jiang, Head of thoracic surgery, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K17-151
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Chemotherapy, Adjuvant; Lung Adenocarcinoma, Stage I; Treatment; Histological Type of Neoplasm
Keywords: Adjuvant chemotherapy; Micropapillary Component; Early stage lung cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Neoplasms by Histologic Type | interventions — Cisplatin; Carboplatin; Pemetrexed; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (Active Comparator): Undergo surgery, followed by observation. Patients receive no further therapy
  Interventions: Procedure: Undergo surgery
- Arm II (Experimental): Undergo surgery, followed by chemotherapy (cis Platinum/Carboplatin, Pemetrexed Disodium). Patients receive chemotherapy comprising cisplatin 75mg/m2 or Carboplatin AUC=5mg/ml/min, and pemetrexed 500mg/m2 in day 1. Treatment continues every 3 weeks for 4 courses.
  Interventions: Drug: cis Platinum/Carboplatin, Pemetrexed Disodium; Procedure: Undergo surgery

INTERVENTIONS:
Drug: cis Platinum/Carboplatin, Pemetrexed Disodium — Intravenous inject Pemetrexed Disodium for Injection over 10 minutes, waiting for at least 30 minutes, then followed by cis Platinum/ Carboplatin over 2 hours
  Other Names: Pemetrexed Disodium for Injection; ALIMTA; Cisplatin; Paraplatin
  Arms: Arm II
Procedure: Undergo surgery — Therapeutic conventional surgery, R0 resection

SUMMARY:
Randomized phase II trial aims to compare surgery with or without adjuvant chemotherapy in treating patients who are pathologically diagnosed as stage I lung adenocarcinoma with micropapillary component no less than 20%.

DETAILED DESCRIPTION:
The presence of micropapillary component in adenocarcinoma is a predictor of poor prognosis, and has been reported to be to be chemosensitive to platinum-based chemotherapy. Seeking a more appropriate treatment for these patients, we perform this randomized phase II clinical trial. About 460 stage I lung adenocarcinoma patients with micropapillary component ≥ 20% will be included and divided into two group. Patients in the control group will only undergo complete R0 resection of the lesion, no further therapy will be used. While patients in the experimental group are going to receive platinum-based chemotherapy (comprising cisplatin and pemetrexed disodium)about 1 month after therapeutic surgery. Treatment continues every 3 weeks for 4 courses. Clinic and telephone follow up will be conducted for survival data monitoring.

DFS(disease free survival rate) and OS(overall survival rate) curves will be calculated using the Kaplan-Meier, life-table method. Comparison of the survival curve for the two groups will be performed using the log-rank test.

ELIGIBILITY:
Inclusion Criteria:

* Completely resected Stage I NSCLC as defined by the International Staging System
* Pathologically diagnosed Stage I micropapillary predominant lung adenocarcinoma
* Patients must be randomized within 4 weeks from the date of surgery
* No prior chemotherapy or radiation for non-small cell lung cancer
* Performance status of 0 or 1
* Women must be non-pregnant and non-lactating; patients of childbearing potential must agree to use an effective form of contraception while on study
* Patients must have no history of previous or concomitant malignancy, other than curatively treated carcinoma in situ of the cervix, or basal cell or squamous cell carcinoma of the skin, or surgically treated in situ carcinoma of the breast, or other cancer for which the patient has been disease free for five years
* Granulocytes >= 1,800/ul
* Platelets >= 100,000/ul
* Bilirubin < 1.5 mg/dl
* SGOT(serum glutamic-oxaloacetic transaminase) (AST) < 2.0 x ULN(upper limit of normal value)

Exclusion Criteria:

* Do not meet the inclusion criteria
* There is evidence of distant metastases
* Suffered from other malignancies in five years
* Within the past January subjects received other drug trials
* Having serious allergies or idiosyncratic persons, such as you can not use folic acid, dexamethasone, vitamin B12 patients
* Severe lung or heart disease, a history
* Refuses or is unable to sign informed consent to participate in trials
* The abuse of drugs or alcohol addicts.
* Patients with difficult to control bacterial, viral, fungal infections
* Having a personality or mental disorders, without civil capacity or restricted civil capacity.
* Being pregnant or lactating women.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Disease-Free-Survival-Rate | up to 60 months
  the percentage of people in the trial who are alive and cancer free after a specified number of years

SECONDARY OUTCOMES:
Overall-Survival-Rate | up to 60 months
  the percentage of people in the trial who alive, with or without signs of cancer
Disease-Free-Survival-Time | up to 60 months
  From date of diagnosis until the date of first documented progression or date of cancer related death , whichever came first
Overall-Survival-Time | up to 60 months
  Time from randomization until death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Thoracic Surgery Department of Shanghai Pulmonary Hospital, Shanghai, China